CLINICAL TRIAL: NCT03041922
Title: Estimation of Changes in Soft Tissue Rigidity of the Buttocks in Sitting Under Weight Bearing Compared to Sitting Without Weight Bearing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, LEONID CHERVINSKY, Radiologist, HaEmek Medical Center, Israel
Other Study IDs: 0026-16-CMC
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Changes in Elasticity Duo to Pressure Ulcers in Buttocks
Keywords: Elastography; Buttocks; Ultrasound; Soft tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy group: Every participant passes one ultrasound exam for soft tissues in buttocks in order to measure the elasticity of soft tissues in sitting and lying down positions. This kind of exam may help to predict a development in pressure ulcers

SUMMARY:
Estimation of Changes in Soft Tissues Elasticity in Buttocks in lying down and sitting positions by using ultrasound device. the elasticity of fat and muscle tissues will be measured.

May ultrasound exam helps to predict the development of pressure ulcers in buttocks due to continuous sitting.

DETAILED DESCRIPTION:
The purpose of the current new research is to check whether Ultrasound device can be used as a tool for assessing the elasticity of the soft tissues in buttocks and measuring the elasticity of these tissues with and without bearing weight on a healthy population to set standards of normal values.

The far purpose of the research is to use ultrasound device for predicting the development of pressure ulcers.

Population and Methods: In this study, Up to 15 healthy people will participate. Each participant will pass ultrasound scans of the buttocks, lying down and sitting on a chair designed for the purpose of research and this after signing an informed consent form.

The process:

1. The participant lies on his stomach on a bed to determine the location of the muscle that will be marked by a marker.By ultrasound, the investigator measures the thickness of fat and muscle tissues between the Ischial Tuberosity (ITs) and the skin.
2. The participant sits without bearing weight on a chair built for this study, the seat is constructed from five straps. Non-weight bearing test is when the straps are far from the test area, the transducer is placed on the marked place, thickness and elasticity of muscle tissue and fat will be measured.
3. The participant sits with bearing weight on the chair. weight bearing test is when the straps are close to the test area , the transducer is placed on the marked place, thickness and elasticity of muscle tissue and fat will be measured.

After measuring the elasticity of the soft tissues,the data will be analyzed in order to define ranges of differences between elasticity with and without weight bearing.

ELIGIBILITY:
Inclusion Criteria: healthy volunteers, BMI- 18.5-29.9,

-

Exclusion Criteria:

* People with neurological deficit
* people with diabetes
* people with a BMI above 29.9 or below 18.5
* pregnant women
* people with bedsores
* mental incompetence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gender: all Age Limits: above 18 years old Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Elasticity values to be measured by ultrasound device | Each exam takes about 30 minutes
  Elastography software in ultrasound device enable to measure the elasticity of soft tissues in human body in kilo pascal units.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Leonid Chervinsky, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: research: The relationship between pressure ulcer incidence and buttock-seat cushion interface pressure in at-risk elderly wheelchair users. — https://www.ncbi.nlm.nih.gov/pubmed/11295017
- See also: research: The effect of mechanical strains in soft tissues of the shoulder during load carriage — https://www.ncbi.nlm.nih.gov/pubmed/26542788